CLINICAL TRIAL: NCT06410040
Title: A Retrospective Study of the Efficacy and Safety of Lolatinib in Anaplastic Lymphoma Kinase (ALK) - Positive Non-Small Cell Lung Cancer (NSCLC) Patients With Brain or Meningeal Metastasis
Brief Title: A Retrospective Study of the Efficacy and Safety of Lolatinib in ALK+ NSCLC Patients With Brain or Meningeal Metastasis
Status: Active, not recruiting | Type: Observational
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Juan LI, MD, Principal Investigator, Sichuan Cancer Hospital and Research Institute
Other Study IDs: EK2023003
Record Dates: First submitted 2024-05-05; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: ALK-positive Non-small Cell Lung Cancer; Brain Metastases; Meningeal Metastasis
MeSH Terms: conditions — Brain Neoplasms; Meningeal Carcinomatosis | interventions — lorlatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced ALK+ NSCLC Patients with Brain or Meningeal Metastasis
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — lolatinib 100mg qd po

SUMMARY:
This study was a retrospective observational study. The study included patients with non-small cell lung cancer with ALK-fusion brain metastases or meningeal metastases who received first-line and late-line treatment with the third-generation ALK TKI lorlatinib between June 2022 and June 2023.

Data were collected from the electronic medical records database and hospital information system of many hospitals in Sichuan Province. Clinical pathology features including gender, age, ALK mutation status at diagnosis, and clinical stage at diagnosis were collected from the medical records. The physical condition assessed by ECOG-PS before the administration of lorlatinib was recorded. Information on anti-tumor therapy was obtained from the records, including dose and time of ALK-TKI therapy and tumor response, number of prior systemic therapy lines, drug regimen, efficacy, and whether local therapy such as radiotherapy and surgery had been received. In this study, the sample size is not limited, and information is collected according to the maximum number of patients. The study period was from 01 July 2023 to 30 June 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosis of advanced NSCLC with clear pathology and brain metastases confirmed by MRI or CT scan of the brain or meningeal metastases confirmed by imaging or lumbar puncture cerebrospinal fluid cytology
3. ALK fusion mutation confirmed by tumor histology or hematology
4. Treatment with lorlatinib from June 2022 to June 2023
5. Survival greater than 12 weeks

Exclusion Criteria:

Patients treated with lorlatinib for less than 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ALK-mutated non-small cell lung cancer patients with brain or meningeal metastasis were included.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | From date of receiving therapy until date of disease progression or the end of study, whichever came first, assessed up to 24 months.
  the Sum of percentage of participants with CR and PR as assessed by RECIST v1.1 or RANO-BM criteria every 8-12 weeks.

SECONDARY OUTCOMES:
PFS | From date of receiving therapy until date of disease progression or death, whichever came first, up to approximately 24 months.
  Intracranial and systemic PFS as assessed by the investigators using RECIST V1.1 or RANO-BM Separately.
OS | From date of receiving therapy until date of disease progression or death, whichever came first, assessed up to approximately 24 months.
  Overall survival for first-line and late-line of lorlatinib medication
AE | From date of receiving therapy until date of disease progression or death or the end of study, assessed up to approximately 24 months.
  Number and percentage of participants with treatment-related AEs as assessed by CTCAE v5.0, and the duration of AEs on every grade

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan cancer hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No